CLINICAL TRIAL: NCT01148407
Title: Platelet Modulation in the Control of Angiogenesis: A Study of Angiogenic and Coagulation Proteins in Patients With Cancer
Brief Title: Platelet Modulation: A Study of Angiogenic and Coagulation Proteins in Patients With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Chris E. Holmes, MD, PhD, University of Vermont
Other Study IDs: VCC 0806
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Cancer
Keywords: breast cancer; platelets; metastatic cancer; malignancy
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — plasma, serum and platelet activated blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood samples on persons with cancer will be sampled for angiogenic, metastatic and coagulation proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of malignancy

Exclusion Criteria:

* Patients taking aspirin, NSAIDs, warfarin or platelet inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a malignancy diagnosis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chris E Holmes, MD PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont/Fletcher Allen Health Care, Burlington, Vermont, United States